CLINICAL TRIAL: NCT07136558
Title: An Open-Label, Multi-center, Phase I Study to Evaluate the Safety, Tolerability, Pharmacokinetics, and Efficacy of ICP-B794 in Patients With Advanced Solid Tumors
Brief Title: Evaluation of ICP-B794 in Patients With Advanced Solid Tumors
Status: Not yet recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Beijing InnoCare Pharma Tech Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ICP-CL-01501
Record Dates: First submitted 2025-08-05; First posted 2025-08-22 (Actual); Last update posted 2025-08-22 (Actual); Status verified 2025-08

CONDITIONS: Advanced Solid Tumors

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- ICP-B794 (Experimental)
  Interventions: Drug: ICP-B794

INTERVENTIONS:
Drug: ICP-B794 — Intravenous administration once every 3 weeks

SUMMARY:
An Open-Label, Multi-center, Phase I Study to Evaluate the Safety, Tolerability, Pharmacokinetics, and Efficacy of ICP-B794 in Patients with Advanced Solid Tumors

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥18 years and ≤75 years.
2. Histologically confirmed other locally advanced or metastatic solid tumors.
3. Life expectancy ≥3 months.
4. Adequate organs function within 7 days prior to the first dose of ICP-B794
5. Eastern Cooperative Oncology Group Performance Status (ECOG PS) score of 0 or 1。
6. At least one measurable lesion per RECIST V1.1 criteria.
7. Able to provide archived tumor tissue sample (within 2 years) or fresh tumor tissue sample.
8. Female participants of childbearing potential (WOCBP) must have a negative serum pregnancy test at screening.
9. WOCBP and male participants must agree to use contraceptive method.
10. Female participants must not breastfeed or plan pregnancy during the study and for at least 6 months after the last dose of investigational drug.
11. Participants must be able to communicate effectively with investigators and comply with all study requirements.
12. Participants voluntarily joined the study and signed the informed concent form (ICF).

Exclusion Criteria:

1. Other active primary malignancies within 3 years prior to the first dose of investigational product.
2. Prior or current treatment with the similar drug or related treatment specified in the protocol.
3. Having a past medical history and unhealthy lifestyle history as specified in the protocol, or suffering from diseases as specified in the protocol.
4. Toxicities from prior anti-tumor therapy not recovered to ≤ Grade 1 (per CTCAE V5.0).
5. Major arterial or venous thrombotic events within 3 months prior to first dose.
6. Active bleeding within 2 months prior to screening or history of clinically significant bleeding tendency.
7. Major surgery within 28 days prior to first dose or minor surgery within 2 weeks prior to first dose.
8. Requirement for systemic corticosteroid therapy within 14 days prior to first dose.
9. History of severe hypersensitivity, or known severe hypersensitivity to the active pharmaceutical ingredient, inactive ingredients in the drug product, or antibody-based drugs, or hypersensitivity to recombinant human or murine proteins, or history of severe infusion reaction.
10. Administration of any live vaccine within 4 weeks prior to first dose or history of hypersensitivity reactions of any grade.
11. Female participants who are pregnant, lactating, or planning pregnancy during the study.
12. Any psychiatric or cognitive disorder that may impair understanding or execution of the informed consent document and/or protocol compliance
13. Other conditions determined by the investigator that render patients unsuitable for participation in this study.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 410 (Estimated)
Dates: Start 2025-08 (Estimated); Primary Completion 2029-06 (Estimated); Study Completion 2030-12 (Estimated)

PRIMARY OUTCOMES:
Incidence, character, and severity of adverse events (AEs) as judged according to NCI-CTCAE v5.0 | Up to 2 years
Dose-limiting toxicities (DLT) | Up to 2 years
  Incidence, character, and severity of dose-limiting toxicities.
The Recommended Dose (RD) of ICP-B794 for expansion and Maximum Tolerated Dose (MTD) | Up to 2 years
Objective response rate (ORR) | Up to 2 years

SECONDARY OUTCOMES:
Maximum Plasma Concentration (Cmax) | Up to 2 years
Time to Maximum Plasma Concentration (Tmax) | Up to 2 years
Half-life (T1/2) | Up to 2 years
Area under the concentration-time curve from zero time to infinity (AUC0-∞) | Up to 2 years
Area under the concentration-time curve from zero time to the last measurable concentration time point t (AUC0-t) | Up to 2 years
Apparent Clearance (CL/F) | Up to 2 years
Terminal Apparent Volume of Distribution (Vz/F) | Up to 2 years
Objective Response Rate (ORR) | Up to 2 years
Disease control rate (DCR) | Up to 2 years
Duration of response (DOR) | Up to 2 years
Progression-Free Survival (PFS) | Up to 2 years
Radiographic progression-free survival (rPFS) | Up to 2 years
Overall survival (OS) | Up to 2 years
Number of participants with anti-drug antibodies (ADA) to ICP-B794 | Up to 2 years

OTHER OUTCOMES:
B7-H3 protein expression | Up to 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Yilong Wu, Principal Investigator — Guangdong Provincial People's Hospital
Locations (1):
- Guangdong Provincial People's Hospital, Guangzhou, Guangdong, China